CLINICAL TRIAL: NCT01618409
Title: PictureRx: An Intervention to Reduce Latino Health Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PictureRx, LLC (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, M Brian Riley, Director of Research, PictureRx, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R43MD004048 (NIH); 5R43MD004048-02 (NIH)
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Medication Adherence; Diabetes
Keywords: PictureRx; Health Literacy; Limited English Proficiency; Latinos; Spanish
MeSH Terms: conditions — Medication Adherence; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PictureRx cards (Experimental): Illustrated format of medication instructions that includes pictures of pills and icons to show their purpose
  Interventions: Behavioral: PictureRx card
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: PictureRx card — An illustrated format of medication instructions that includes pictures of the medications and icons to illustrate their purpose
  Arms: PictureRx cards

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the effect of Spanish-language illustrated medication instructions (PictureRx cards), compared to traditional medication instructions, on Latinos' understanding of their medication regimens. The study will also assess the effect on self-reported medication adherence. Patients with diabetes who attend participating clinics are eligible. The target sample size is 200.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Latino, Spanish speaker
* Be at least 18 years old
* Must be taking at least 1 chronic medication

Exclusion Criteria:

* Too ill to participate in an interview
* Do not have a telephone
* Having visual acuity worse than 20/50 via Rosenbaum Visual Acuity exam (eyechart)
* Inability to communicate in either Spanish or English
* Overt psychiatric illnesses, overt delirium or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Patient Understanding of their Medication Regimen | Approximately 1 week after enrollment
  The primary outcome will be patients' understanding of their medication regimen, as assessed by an interviewer-administered questionnaire.

SECONDARY OUTCOMES:
Self-reported Adherence | Approximately 1 week after enrollment
  As a secondary outcome, patients will report their self-reported adherence using a validated instrument.

CONTACTS AND LOCATIONS:
Overall Officials: M Brian Riley, MA, Principal Investigator — PictureRx, LLC
Locations (1):
- Saint Thomas Family Health Center - South, Nashville, Tennessee, United States